CLINICAL TRIAL: NCT02512692
Title: A Traditional Feasibility Study of Gemcitabine, Cisplatin, and 90Y TARE for Unresectable Intrahepatic Cholangiocarcinoma
Brief Title: Gemcitabine-Cisplatin-90Y TARE for Unresectable Intrahepatic Cholangiocarcinoma
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrollment closed by internal scientific review committee due to slow accrual.
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 102254
Record Dates: First submitted 2015-07-29; First posted 2015-07-31 (Estimated); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Intrahepatic Cholangiocarcinoma
Keywords: intrahepatic cholangiocarcinoma; cholangiocarcinoma; 90Y TARE; radioembolization; gemcitabine and cisplatin
MeSH Terms: conditions — Cholangiocarcinoma | interventions — Gemcitabine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: Yes

ARMS (1):
- 90Y TARE with Gemcitabine and Cisplatin (Experimental): 90Y TARE will be given on day 3 or 4 of cycle 1 and start at 75% of the dose calculated by the body surface area formula and escalated by 25% per cohort in combination with cisplatin 25 mg/m2 and gemcitabine 300 mg/m2 in cycles 1 and 2.
  Once the 90Y TARE has reached the 100% dose level, the gemcitabine dose will increase to 600mg/m2 in dose level 3 and 1000mg/m2 in dose level 4. The cisplatin dose will remain at 25/mg/m2.
  For all dose levels, from cycle 3 to cycle 8, the cisplatin dose will be 25mg/m2 and the gemcitabine dose will be 1000mg/m2.
  Interventions: Device: SIR-Spheres microspheres (Yttrium-90 Microspheres); Drug: Gemcitabine; Drug: Cisplatin

INTERVENTIONS:
Device: SIR-Spheres microspheres (Yttrium-90 Microspheres) — On Day 3 or 4 of cycle 1 90Y TARE will be administered
  Other Names: 90Y TARE
Drug: Gemcitabine — On days 1 and 8 of each cycle (21 days) Gemcitabine will be administered. Treatment may last up to 8 cycles
Drug: Cisplatin — On days 1 and 8 of each cycle (21 days) Cisplatin will be administered. Treatment may last up to 8 cycles

SUMMARY:
The purpose of this study is to determine the safety and maximum tolerated dose (MTD) of 90 Y TARE (Y90) in combination with gemcitabine and cisplatin in patients with unresectable intrahepatic cholangiocarcinoma (ICC).

DETAILED DESCRIPTION:
Gemcitabine and cisplatin chemotherapy is the current standard for the treatment of unresectable intrahepatic cholangiocarcinoma. 90Y TARE combined with the current standard may be an ideal way to improve disease control in the liver as almost all patients die from their disease in the liver. The data from this trial would then be used to move to a phase II trial to determine efficacy to see if a phase III trial would be warranted. In addition, assessment of the molecular classification of intrahepatic cholangiocarcinoma could determine if there is difference in survival with chemotherapy and 90Y TARE. Finally, MRI before and after treatment will be used to determine if utilizing the percent increase of mean ADC correlates with survival.

ELIGIBILITY:
Inclusion Criteria:

* Histologic Documentation: Core needle biopsy or surgical specimen that confirms intrahepatic cholangiocarcinoma (ICC). Patients must be determined to be unresectable by a multidisciplinary team that includes a hepatobiliary surgeon.
* No prior liver radiation therapy or immunotherapy for cholangiocarcinoma.
* Only one previous single agent chemotherapy for ICC allowed.
* Patient may have prior liver resection.
* Age > 18 years of age.
* Eastern Cooperative Oncology Group (ECOG) performance status < 2 (see Appendix E)
* Child's Pugh score of A (see Appendix F)
* Life expectancy of greater than 4 months
* Normal organ and marrow function as outlined in the protocol.
* Willingness to use effective contraceptive methods during the study. Patient may participate in the female (or female partner of male subject), either is not of childbearing potential (defined as postmenopausal for > 1 year or surgically sterile) or is practicing two forms of contraception. Sexually active male participants must agree to use a physical barrier method (male latex rubber condom with or without spermicide).
* Patients with well controlled HIV infection are eligible if their CD4 count is >499/cu mm and viral load is < 50 copies/ml.
* Pre-certification for the 90Y TARE should be performed prior to enrollment on this study.
* All patients must be informed of the investigational nature of this study and must have the ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients who have had major surgery within 4 weeks prior to entering the study or those who have not recovered from complications from a surgery more than 4 weeks earlier.
* Patients may not be receiving any other investigational agents.
* Patients must not have any grade III/IV cardiac disease as defined by the New York Heart Association (NYHA) Criteria
* Patients must NOT have liver disease such as cirrhosis or sever hepatic impairment as defined by Child-Pugh Class B or C
* Pregnant women are excluded from this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2015-07-21 (Actual); Primary Completion 2021-03-19 (Actual); Study Completion 2021-03-19 (Actual)

PRIMARY OUTCOMES:
To determine the feasibility of 90Y TARE in combination with gemcitabine and cisplatin in patients with unresectable intrahepatic cholangiocarcinoma. | Up to 2 years
  A continual reassessment method (CRM) design will be used to confirm the Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 in regards to 90Y TARE.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel L. Cooper, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-11-14): https://cdn.clinicaltrials.gov/large-docs/92/NCT02512692/Prot_SAP_000.pdf
  • Informed Consent Form (2016-07-19): https://cdn.clinicaltrials.gov/large-docs/92/NCT02512692/ICF_001.pdf